CLINICAL TRIAL: NCT00449462
Title: The Effect of Conjugated Linoleic Acid Intake on Liver and Kidney Function in Healthy Volunteers (CLAxon-Study)
Brief Title: Effect of Conjugated Linoleic Acid Intake on Liver and Kidney Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: VU University of Amsterdam (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL15420.081.06
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-03

CONDITIONS: Healthy
Keywords: CLA; liver; kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: consumption of CLA enriched food

SUMMARY:
The knowledge of the health effects of CLA on the human body is limited. However, CLA supplements are sold over the counter in several countries and various techniques are used to increase the content of CLA in food.

The CLAxon-study will be performed to investigate wether high doses of CLA can be safely given to healthy human volunteers.

DETAILED DESCRIPTION:
Each volunteer receives CLA enriched products for a total of 3 weeks containing approximately 20g CLA per day. A control group is not needed. If three subjects or more show one or more blood values for liver and kidney function above predefined limits the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* serum total cholesterol < 8.0 mmol/L
* serum triglycerides < 3.0 mmol/L
* ALAT < 45 IU/L
* ASAT < 41 IU/L
* amylase 35-130 U/L
* alkaline phosphatase 40-125 U/L
* bilirubin < 17 µmol/L
* gamma-glutamyltranspeptidase > 75 U/L (men) and < 40 U/L (women)
* lactate dehydrogenase 230-485 U/L
* creatinine clearance >= 90 mL/min
* fasting glucose levels 70-115 mg/dL
* fasting insulin levels 5-30 mU/L

Exclusion Criteria:

* use of cholesterol lowering medication
* high alcohol intake
* BMI > 30
* chronic diseases (such as diabetes, cardiovascular disease, kidney and liver dysfunction)
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
ALAT
ASAT
amylase
bilirubin
alkaline phosphatase
gamma-glutamyltranspeptidase
lactate dehydrogenase
creatinine clearance

SECONDARY OUTCOMES:
total cholesterol
HDL cholesterol
LDL cholesterol
triglycerides
fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg A Brouwer, PhD, Principal Investigator — VU University of Amsterdam; Martijn B Katan, Professor, Principal Investigator — VU University of Amsterdam
Locations (2):
- Netherlands (2):
  - VU University Amsterdam, Institute for Health Sciences, Amsterdam
  - Wageningen University, Division of Human Nutrition, Wageningen

REFERENCES:
- [Derived] Wanders AJ, Leder L, Banga JD, Katan MB, Brouwer IA. A high intake of conjugated linoleic acid does not affect liver and kidney function tests in healthy human subjects. Food Chem Toxicol. 2010 Feb;48(2):587-90. doi: 10.1016/j.fct.2009.11.036. Epub 2009 Nov 22. PMID 19932729